CLINICAL TRIAL: NCT02673359
Title: Vaginal Progesterone Versus Cervical Cerclage for Pregnant Women With Sonographic Short Cervix and History of Preterm Labor and/or Midtrimester Miscarriage
Brief Title: Vaginal Progesterone Versus Cervical Cerclage for Pregnant Women With Short Cervix and History of PTL and/or MTM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WR2
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Premature Labour
Keywords: Preterm labor; Short cervix; Progesterone; Cervical cerclage
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone; Cerclage, Cervical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone group (Active Comparator): Vaginal progesterone suppositories will be given
  Interventions: Drug: Progesterone
- Cerclage group (Active Comparator): Cervical cerclage will be performed.
  Interventions: Procedure: Cervical cerclage

INTERVENTIONS:
Drug: Progesterone — Vaginal progesterone suppositories (Cyclogest®, Actavis, Barnstaple, EX32 8NS, United Kingdom) will be given in a dose of 400 mg/day
  Other Names: Cyclogest; Prontogest
  Arms: Progesterone group
Procedure: Cervical cerclage — Cervical cerclage will be performed by transvaginal placement of purse-string stitch suture at the cervicovaginal junction, without mobilization of the urinary bladder (McDonald cervical cerclage)
  Other Names: Cervical stitch
  Arms: Cerclage group

SUMMARY:
The aim of this study to compare vaginal progesterone supplementation to cervical cerclage for prevention of preterm labor in women with short cervical length and history of previous midtrimester miscarriage and/or preterm labor.

DETAILED DESCRIPTION:
Women with singleton pregnancy and history of preterm labor and/or midtrimester miscarriage in a previous pregnancy will be selected for serial assessment of the cervical length by transvaginal sonography (TVS) starting from 16 weeks till 24 weeks of gestation. Eligible participants in our study will be those who have cervical length of 15-25 mm at 16-24 weeks of gestation. At 16-24 weeks gestational age, all women participating in the study will be randomly allocated into two groups; progesterone group and cerclage group. For women in the progesterone group, vaginal progesterone suppositories will be given in a dose of 400 mg/day. For women in the cerclage group, McDonald cervical cerclage will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy.
* History of preterm labor and/or midtrimester miscarriage in a previous pregnancy.
* Cervical length of 15-25 mm by transvaginal sonography (TVS) at 16-24 weeks of gestation.

Exclusion Criteria:

* Age < 20 or > 35 years.
* Congenital uterine malformation.
* Multifetal pregnancy.
* Known major fetal structural or chromosomal abnormality.
* Known allergy or contraindication (relative or absolute) to progesterone therapy.
* Presence of contraindication to cervical cerclage.
* Medical conditions complicating pregnancy.
* Vaginal bleeding.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-02; Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Preterm labor before 35 weeks | Up to 35 weeks gestational age

SECONDARY OUTCOMES:
Delivery before 37 weeks | Up to 37 weeks gestational age
Low birth weight (LBW) | At birth
  Birth weight of a living neonate of < 2500 gm regardless of gestational age
Neonatal respiratory distress syndrome (RDS) | At birth
Early neonatal death (END) | One month after birth

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-refaie, Dr, Principal Investigator — Port Said University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University; Ahmed M Badawy, Prof, Study Chair — Mansoura University
Locations (3):
- Egypt (3):
  - Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private practice settings, Al Mansurah, Dakahlia Governorate
  - Obstetrics and Gynecology Department in Port Said University, Port Said

IPD SHARING:
Plan to Share IPD: Undecided